CLINICAL TRIAL: NCT04538768
Title: Prevention of Lateral Incisional Hernia After Stomal Closure Using P4HB Retro-muscular Mesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Buccheri La Ferla Hospital, Palermo (Other)
Responsible Party: Principal Investigator, Leo Licari, Principal Investigator, Buccheri La Ferla Hospital, Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20082020
Record Dates: First submitted 2020-08-22; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Incisional LLQ Hernia
Keywords: lateral incisional hernia; mesh augmentation; prevention; stomal closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesh Augmentated (Experimental)
  Interventions: Procedure: Mesh augmentation
- Direct Suture (Other)
  Interventions: Procedure: Direct suture

INTERVENTIONS:
Procedure: Mesh augmentation — P4HB retromuscular mesh placement for prevention of lateral incisional hernia after stomal closure
  Arms: Mesh Augmentated
Procedure: Direct suture — direct fascia suture
  Arms: Direct Suture

SUMMARY:
The aim of the study is to determine whether the use of the P4HB retro muscular mesh can prevent the lateral incisional hernia after stomal closure.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 y.o.
* stomal closure
* elective surgery

Exclusion Criteria:

* patients < 18 y.o.
* emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
rate of postoperative lateral incisional hernia after P4HB mesh placement vs direct fascia suture. | 1 week to 18 months after surgery
  the outcome 1 will be assessed through clinical examination during follow up time. when the suspicion of incisional hernia will be hypothesized the patients will be conducted to perform US of the abdomen and CT scan of the abdomen if strictly required to confirm the suspicion.

SECONDARY OUTCOMES:
surgical operation time in P4HB mesh placement group vs direct fascia suture group. | intraoperative
  outcome 2 will be assessed through the measurement of the length of surgical operation. The length of the surgical operation will be measured in minutes from the incision of the skin to the suture of the skin. data will be compared with those of the control arm (direct fascia suture) to understand the feasibility of the technique proposed.
length of hospital stay in P4HB mesh placement group vs direct fascia suture group. | From the starting date of the study until the date of its completion, assessed up to 18 months"
  outcome 3 will be assessed through the measurement of the length of the hospital stay. The length of hospital stay will be measured in days from admission to dimission of the patient. Data will be compared with those of the control arm (direct fascia suture).
rate of surgical site infection in P4HB mesh placement group vs direct fascia suture group. | 1 week after surgery; 1 month after surgery; 3 months after surgery; 6 months after surgery; 12 months after surgery; 18 months after surgery
  outcome 4 will be assessed through clinical examination during follow up time evaluating the rate of postoperative complication such as surgical site infection.
rate of seroma formation in P4HB mesh placement group vs direct fascia suture group. | 1 week after surgery; 1 month after surgery; 3 months after surgery; 6 months after surgery; 12 months after surgery; 18 months after surgery
  outcome 5 will be assessed through clinical examination during follow up time evaluating the rate of postoperative complications such as seroma.
rate of hematoma formation in P4HB mesh placement group vs direct fascia suture group. | 1 week after surgery; 1 month after surgery; 3 months after surgery; 6 months after surgery; 12 months after surgery; 18 months after surgery
  outcome 6 will be assessed through clinical examination during follow up time evaluating the rate of postoperative complications such as hematoma.
assessment of quality of life (QoL) through QoL scale in P4HB mesh placement group vs direct fascia suture group. | 18 months after surgery.
  outcome 7 will be assessed through assessment of the postoperative QoL. The SF-36 questionnaire will be administered post-operatively.
  The 36-Item Short Form Health Survey questionnaire (SF-36) is a very popular instrument for evaluating Health-Related Quality of Life.
  The SF-36, as described in the name, is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
cost effectiveness analysis of the P4HB mesh augmentation technique vs direct fascia suture group. | through study completion, an average of 1 year .
  the outcome 8 will be assessed through the collection of data about the total costs for the surgical operation and the hospitalization considering materials and mesh used. The analysis will be used to compare the costs of the technique proposed with those of the incisional hernia management in order to conduct a cost effectiveness analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Leo Licari, MD, Study Director — Ospedale Buccheri La Ferla Palermo; University of Palermo - Department of Surgical, Oncological and Oral Sciences; Cosimo Callari, MD, Study Chair — Ospedale Buccheri La Ferla Palermo
Locations (1):
- Ospedale Buccheri La Ferla Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes